CLINICAL TRIAL: NCT06220747
Title: Effectiveness of Single Dose or Two Doses of HPV Vaccine Among Adolescents and Reproductive Women: A Test-negative Control Study
Brief Title: Effectiveness of HPV Vaccine Among Adolescents and Reproductive Women
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor Emeritus, Mahidol University
Other Study IDs: NRCT9-3
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hpv
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — urine collection 10-30 ml. and self cervical swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women aged 12-45 years old

SUMMARY:
To assess the effectiveness of HPV vaccine 2 doses or less to prevent HPV high risk infection among adolescents and adults. We conduct the test-negative control study including 12-45 women who interest to do a check-up pap smear. Cases were women who met the inclusion criteria and tested positive for HPV DNA, and controls were defined as women who met inclusion criteria but tested negative. For the proposed HPV VE study, we will enroll nine controls for each enrolled case. The participants will be interviewed about their demographics and vaccine histories. Potential confounders data will be collected by interview or self- report questionnaire. HPV DNA test will be done by urine or self-cervical sampling (optional). In case the participant has previous HPV test result within 1 year, the result will be recorded and analysed without repeating the test.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 12-45 who willing to do HPV test check-up.
* Subject has provided written informed consent prior to performance of any study-specific procedures and is willing and has means to be contacted and to contact the investigator during the study.
* Based on clinical judgment, the participant with underlying chronic disease who has stable and well-controlled medical conditions.

Exclusion Criteria:

* Participant with history of total hysterectomy and loop electrosurgical excision procedure.
* Participant who received 3 doses HPV vaccine.
* Any condition that might confound the interpretation of vaccine effectiveness by investigator

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Target populations are any women aged 12-45-year-old who interest this project.
  For the proposed HPV VE study, we will enroll nine controls for each enrolled case. The participants will selection based on their outcome, not based on exposure. Cases were women who met the inclusion criteria and tested positive for HPV DNA (self-cervical swab/ urine sample: positive), and controls were defined as women who met inclusion criteria but HPV DNA tested negative.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The real world effectiveness of HPV vaccine 2 doses or less to prevent HPV high risk infection among women aged 12-45 | 1 visit (1 day)
  Estimation of overall vaccine effectiveness For the planned analyses, the log odds of disease for individuals in matched sets will be modelled using the following conditional logistic model:Model 1 : Log (oddcase) = α¬i + β e(HPV_vaccination) + β1(cov_1) +β2(cov_2) + ... + βk(cov_k)where αi is the stratum-specific constant term for each matched set, βe is the parameter coefficient for the exposure of interest (receipt of HPV vaccine), and β1 through βk are the parameter coefficients for each covariate included in the model to control for confounding. Our modelling strategy will be to create models that always contain the exposure variable of interest (receipt of HPV vaccine) and additional covariates as needed.

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Prof., Study Chair — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University
Locations (2):
- Thailand (2):
  - Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok, Select...
  - Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, 420/6 Ratchawithi Road, Ratchathewi,, Bangkok